CLINICAL TRIAL: NCT03109756
Title: A Phase 1 Single Dose PK Study in Adolescent Subjects With Fragile X Syndrome or Angelman Syndrome
Brief Title: Single Dose Pharmacokinetic (PK) Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Healx AI (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OV101-16-001
Record Dates: First submitted 2017-04-06; First posted 2017-04-12 (Actual); Last update posted 2017-11-30 (Actual); Status verified 2017-09

CONDITIONS: Angelman Syndrome; Fragile X Syndrome
MeSH Terms: conditions — Angelman Syndrome; Fragile X Syndrome | interventions — gaboxadol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Single-dose 5 mg OV101 (Experimental)
  Interventions: Drug: OV101

INTERVENTIONS:
Drug: OV101 — Single-dose 5 mg OV101
  Other Names: Gaboxadol

SUMMARY:
The trial is a Phase 1 Single Dose PK Study in Adolescent Subjects with Fragile X syndrome (FXS) or Angelman syndrome (AS).

* The primary objective of the study is to evaluate the pharmacokinetics (PK) of OV101 following a single 5 mg dose of OV101 in adolescents with FXS or AS.
* Secondary objectives are to determine the safety and tolerability of a single 5 mg dose of OV101 in adolescents with FXS or AS.

ELIGIBILITY:
Inclusion Criteria:

1. Adolescents with confirmed clinical and previous molecular diagnosis of FXS or AS, age between 13 to 17 years, inclusive.
2. Subjects must assent to participation in the study (if appropriate), have a parent or legal guardian/representative capable of providing informed consent on behalf of the subject, and commit to participate in all assessments described in the protocol.
3. Subjects must be receiving a stable dose of concomitant medications
4. Subjects should be able to complete study assessments.
5. Subjects who are non-sterile must agree to either remain completely abstinent or to use two effective contraceptive methods from screening until 7 days after the last dose of study treatment.
6. Subjects must have a parent or other reliable caregiver who agrees to accompany the subject at all study visits and provide information about the subject as required by the study protocol, and ensure compliance with the protocol.

Exclusion Criteria:

1. Inability to swallow a capsule.
2. Poorly controlled seizures
3. Clinically significant abnormal ECG at the time of screening.
4. Positive result on serum or urine pregnancy test for women of child-bearing potential (have experienced menarche) who are not using a dual method of contraception (e.g., condoms plus oral contraceptives), with abstinence being an accepted method.
5. Allergy to gaboxadol or any excipients
6. Concomitant cardiovascular, respiratory, liver, renal, or hematologic diseases of a degree that would limit participation in the study
7. History of suicidal behavior or considered a high suicidal risk by the investigator.
8. Any medical, psychological, social disorder(s), or other conditions - including seizure disorder

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 12 (Actual)
Dates: Start 2017-04-03 (Actual); Primary Completion 2017-11-28 (Actual); Study Completion 2017-11-28 (Actual)

PRIMARY OUTCOMES:
Measurement of maximum plasma concentration achieved following a single dose of OV101 | 10 hours
  Maximum plasma concentration (Cmax)
Measurement of time of maximum plasma concentration following a single dose of OV101 | 10 hours
  Time after administration of drug when maximum plasma concentration is reached (Tmax)
Measurement of plasma half-life following a single dose of OV101 | 10 hours
  Plasma half-life (T1/2)
Measurement of the area under the plasma concentration versus time curve following a single dose of OV101 | 10 hours
  Area under the curve from 0 to 10 hours (AUC 0-10)
Measurement of clearance following a single dose of OV101 | 10 hours
  Total body clearance (CL)
Measurement of the apparent volume of distribution following a single dose of OV101 | 10 hours
  Apparent volume of distribution during terminal phase (Vz)

SECONDARY OUTCOMES:
Safety parameters, adverse events, absolute values and changes over time of hematology, clinical chemistry, urinalysis, vital signs, electrocardiogram (ECG) | 10 hours

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Ovid Therapeutics Investigative Site, Chicago, Illinois
  - Ovid Therapeutics Investigative Site, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: No